CLINICAL TRIAL: NCT01343914
Title: Retrospective Study to Determinate the Clinical Phenotype of Patients With Non Squamous NSCLC Treated With First Line Bevacizumab-based Therapy That Reached a Long PFS
Brief Title: An Observational Study on Patients With Non-Squamous NSCLC Who Reached A Long PFS After Avastin (Bevacizumab)-Based First-Line Therapy
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25494
Record Dates: First submitted 2011-04-12; First posted 2011-04-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This retrospective observational study will analyse demographic, clinical and treatment-related data of patients with non-squamous non-small cell lung cancer (NSCLC) who had reached >/= 9 months of progression-free survival after Avastin (bevacizumab)-based first-line therapy. Data will be collected for approximately 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Non-squamous non-small cell lung cancer (NSCLC) treated with first-line Avastin-based therapy
* Progression-free survival of >/= 9 months reached

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non squamous NSCLC patients treated with bevacizumab-based first line therapy and PFS >/= 9 months
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (>9 months) according to clinical phenotype | approximately 9 months

SECONDARY OUTCOMES:
Overall survival | approximately 9 months
Safety: Incidence of adverse events | approximately 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- Spain (23):
  - Alcoy, Alicante
  - Alicante, Alicante
  - Elche, Alicante
  - Elda, Alicante
  - Almería, Almeria
  - Manacor, Balearic Islands
  - Palma de Mallorca, Balearic Islands
  - Barcelona, Barcelona
  - Cáceres, Caceres
  - San Sebastián de los Reyes, Guipuzcoa
  - Jaén, Jaen
  - Santiago de Compostela, La Coruña
  - León, Leon
  - Lugo, Lugo
  - Madrid, Madrid
  - Málaga, Malaga
  - Murcia, Murcia
  - Navarra, Navarre
  - Pontevedra, Pontevedra
  - Vigo, Pontevedra
  - Seville, Sevilla
  - Valencia, Valencia
  - Zaragoza, Zaragoza